CLINICAL TRIAL: NCT06871605
Title: Comparison of Ultrasound-guided Transversalis Fascia Plane Block With Ultrasound-guided Ilioinguinal and Iliohypogastric Nerve Block in the Treatment of Chronic Post-herniorrhaphy Inguinal Pain
Brief Title: Transversalis Fascia Plane vs Ilioinguinal and Iliohypogastric Nerve Block for the Treatment of CPIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TFP vs II-IH for CPIP
Record Dates: First submitted 2025-02-11; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Inguinal Hernia; Groin Hernia
Keywords: Ultrasonography; Ilioinguinal and iliohypogastric nerve; Transversalis Fascia Plane Block
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversalis fascia plane block group (Active Comparator): transversalis fascia plane block for chronic postherniorrhaphy inguinal pain
  Interventions: Procedure: ultrasound-guided transversalis fascia plane block
- ilioinguinal and iliohypogastric nerve block group (Active Comparator): ilioinguinal and iliohypogastric nerve block for chronic postherniorrhaphy inguinal pain
  Interventions: Procedure: ultrasound-guided ilioinguinal and iliohypogastric nerve block group

INTERVENTIONS:
Procedure: ultrasound-guided transversalis fascia plane block — With the patient in the lateral decubitus position, an 8-12 Hz linear ultrasound (US) probe is placed transversely over the iliac crest. The external oblique (EO), internal oblique (IO) and transversus abdominis (TA) muscles are identified so that the abdominal muscles are in the field of view. The TA muscle is then advanced posteriorly until it tapers to the thoracolumbar fascia with its aponeurosis adjacent to the quadratus lumborum (QL) muscle. The 22 gauge block needle is advanced in plane with the US probe. After placing the needle tip in the virtual triangular plane between the posterior edge of the TA muscle, the QL and the underlying transversalis fascia, 4 mL of 0.5% bupivacaine + 2 mL of a total of 8 mg dexamethasone + 4 mL of saline are injected for a total volume of 10 mL.
  Arms: transversalis fascia plane block group
Procedure: ultrasound-guided ilioinguinal and iliohypogastric nerve block group — With the patient in the supine position, an 8-12 Hz linear ultrasound (US) probe is placed medial and cephalal to the anterior superior iliac spine (ASIS), transversely between the ASIS and the umbilicus. The external oblique (EO), internal oblique (IO) and transversus abdominis (TA) muscles are identified so that the abdominal muscles are in the field of view. The II-IH nerves are hyperechogenic in the fascial plane between the IO and TA muscles. A 22 gauge block needle is advanced in plane with the US probe. When the needle tip is advanced to the II and IH nerves, 4 mL of 0.5% bupivacaine + 2 mL total 8 mg dexamethasone + 4 mL saline is injected for a total volume of 10 mL.
  Arms: ilioinguinal and iliohypogastric nerve block group

SUMMARY:
The aim of this study was to compare the efficacy of ultrasound (US)-guided transversalis fascia plane block (TFP) and ilioinguinal (II) and iliohypogastric (IH) nerve block in the treatment of chronic post-herniorrhaphy inguinal pain (CPIP) refractory to conservative treatments. For this evaluation, a numerical rating scale (NRS) will be used before and after both interventions.

DETAILED DESCRIPTION:
Chronic post-herniorrhaphy inguinal pain (CPIP) after inguinal hernia surgery significantly affects quality of life and daily activities. The incidence of this condition ranges from 15% to 53% and its management is often challenging. CPIP is defined as pain lasting more than three months and can be diagnosed if no organic cause can be found to explain the pain at the end of this period. There are various methods in the treatment of CPIP, including medical therapy, nerve blocks and surgical intervention.

The inguinal region is mainly innervated by the ilioinguinal (II) and iliohypogastric (IH) nerves. These nerves are the most commonly damaged structures after inguinal hernia surgery.

However, the II and IH nerves can be easily blocked in isolation throughout their entire course in the groin area or in the abdominal wall at different injection sites using fascial plane blocks such as transversalis fascia plan block (TFP). These blocks are frequently preferred because of their ease of application and wide analgesic effects. Therefore, studies investigating the efficacy of fascial blocks that provide ease of application are increasing.

Although TFP and II-IH blocks have been used in the treatment of acute postoperative inguinal pain, they have been used in a limited number of studies for CPIP; however, no study has compared the efficacy and advers effect rates of these methods.

The primary aim of this study is to compare the efficacy of these two treatment modalities. The secondary aim is to determine the incidence of adverse events associated with US-guided TFP and II-IH nerve block therapy. A total of at least 80 patients will be enrolled for comparison, 40 patients in each group. The NRS score will be compared both within and between groups before, 1 month after and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Complaints of inguinal pain >12 weeks post-herniorrhaphy surgery
* >18 years of age
* Failure of conservative pain management

Exclusion Criteria:

* Other causes of inguinal pain (haematoma, infection, tubo-ovarian disease, abscess, etc., gynaecological, urological and organic pathologies after inguinal hernia, etc.)
* Pregnancy
* Coagulopathy, antiaggregant/anticoagulant/antiplatelet use
* Unstable psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | Change from baseline to 1st and 3rd month after treatment
  NRS is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

SECONDARY OUTCOMES:
procedure-related adverse events | Change from baseline to 1st and 3rd month after treatment
  Any adverse events that occur during and after the TFP and II-IH block procedures will be recorded.
patient satisfaction likert scale | Change from baseline to 30 minutes after procedure
  Patient satisfaction is measured using a five-point Likert scale (1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied and 5 = very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Gevher Rabia Genc Perdecioğlu, Study Chair — Diskapi TRH
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)